CLINICAL TRIAL: NCT05280977
Title: Comparative Effects Of Post Isometric Relaxation And Post Facilitation Stretching On Range Of Motion, Pain And Functional Limitations In Patients With Erector Spinae Tightness: A Randomized Controlled Trial
Brief Title: Effects Of Post Isometric Relaxation And Post Facilitation Stretching On ROM, Pain And Functional Limitations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/1027/2021
Record Dates: First submitted 2022-03-05; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Erector Spinae Tightness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be single blinded as the assessor will be unaware of the treatment that will be given to both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POST ISOMETRIC RELAXATION (Experimental)
  Interventions: Other: POST ISOMETRIC RELAXATION
- POST FACILITATION STRETCHING (Experimental)
  Interventions: Other: POST FACILITATION STRETCHING

INTERVENTIONS:
Other: POST ISOMETRIC RELAXATION — Group A (Post Isometric Relaxation + Conventional Physiotherapy): This group will receive Muscle Energy Technique in addition to conventional physiotherapy for the treatment of erector spinae tightness. The treatment will be given on alternate days for four weeks with 8 - 10 repetitions of METs per session.
  Arms: POST ISOMETRIC RELAXATION
Other: POST FACILITATION STRETCHING — Group B (Post Facilitation Stretching + Conventional Physiotherapy):
  This group will receive Post Facilitation Stretching Technique in addition to conventional physiotherapy for the treatment of erector spinae tightness. The treatment will be given on alternate days for four weeks with 8 - 10 repetitions of METs per session.
  Arms: POST FACILITATION STRETCHING

SUMMARY:
Study Design: Randomized Controlled Trial treatment techniques: post isometric relaxation and post facilitation stretching technique sample size: 35 in each group single blinded Before giving either treatment to each group, baseline data will be collected from each participant and then after 4th week of treatment.

DETAILED DESCRIPTION:
To compare the effects of post isometric relaxation and post facilitation stretching on Rom, pain and functional disability in patients with erector spinae tightness.Study Setting: Bahria International Hospital, Lahore Data will be analyzed using SPSS version 26.The quantitative variables like range of motion will be presented in the form of mean ±SD and qualitative variables like pain and functional disability will be presented in the form of frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* • Pain in lower back for atleast 4 weeks but less than 1 year.

  * Pain relieved by rest.
  * Decreased flexion, extension and lateral flexion of lumbar spine.
  * Individuals having no signs of nerve root irritation (dermatomal pain and paresthesia) and nerve root compression (dermatomal sensory loss, myotomal weakness, loss of reflex)
  * Age group: 30 - 45 years
  * Both male and female

Exclusion Criteria:

* Individuals having other lumbar pathologies like disc problems, ligamentous strains, sciatica etc
* Individuals having any inflammation and malignancy.
* Pregnancy
* Individuals having recent trauma, fracture, or surgery

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-04-02 (Estimated); Study Completion 2022-04-11 (Estimated)

PRIMARY OUTCOMES:
goniometer | 4 WEEKS
  Range of motion will be measured by using universal standard goniometer.The goniometer comprises a body (rotation axis) with two arms attached to it, one being fixed and the other movable. The measurement of the ROM is performed by direct reading of the angle between the axis of rotation at the end of the active ROM of the movement assessed.

SECONDARY OUTCOMES:
visual analog scale | 4 WEEKS
  The Visual Analogue Scale (VAS) is an instrument for the measurement of subjective characteristics or attitudes that cannot be measured directly. It consists of a horizontal line with markings from 0 - 10 where "0" represents "no pain" and "10" represents "worst pain possible". The patient is asked to mark the number on the scale which best describes the level of his/her pain.

OTHER OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 4 WEEKS
  The Oswestry Low Back Pain Disability Questionnaire is designed to assess the level of functional limitations or disability in activities of daily living of the patients with acute or chronic low back pain. It gives subjective percentage score. The questionnaire consists of 10 questions each having 6 options. Each option carries from 0-5 marks in descending order. The total score of the questionnaire is 50 while the minimum score is 0. The patient is asked to fill the questionnaire and their level of disability is assessed by scoring in the end. Their attained score is divided by the total score i-e 50 and is then divided by 100 to get the percentage

CONTACTS AND LOCATIONS:
Overall Officials: SYEDA RAHAT JABEEN, MSPT, Principal Investigator — University of Lahore
Locations (1):
- Bahria International Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Bogduk N. Functional anatomy of the spine. Handb Clin Neurol. 2016;136:675-88. doi: 10.1016/B978-0-444-53486-6.00032-6. PMID 27430435
- [Background] Panjabi MM, Goel V, Oxland T, Takata K, Duranceau J, Krag M, Price M. Human lumbar vertebrae. Quantitative three-dimensional anatomy. Spine (Phila Pa 1976). 1992 Mar;17(3):299-306. doi: 10.1097/00007632-199203000-00010. PMID 1566168
- [Background] Sung PS, Lammers AR, Danial P. Different parts of erector spinae muscle fatigability in subjects with and without low back pain. Spine J. 2009 Feb;9(2):115-20. doi: 10.1016/j.spinee.2007.11.011. Epub 2008 Feb 14. PMID 18280212
- [Background] Friberg O. Clinical symptoms and biomechanics of lumbar spine and hip joint in leg length inequality. Spine (Phila Pa 1976). 1983 Sep;8(6):643-51. doi: 10.1097/00007632-198309000-00010. PMID 6228021
- [Background] Allegri M, Montella S, Salici F, Valente A, Marchesini M, Compagnone C, Baciarello M, Manferdini ME, Fanelli G. Mechanisms of low back pain: a guide for diagnosis and therapy. F1000Res. 2016 Jun 28;5:F1000 Faculty Rev-1530. doi: 10.12688/f1000research.8105.2. eCollection 2016. PMID 27408698
- [Background] Wilson E, Payton O, Donegan-Shoaf L, Dec K. Muscle energy technique in patients with acute low back pain: a pilot clinical trial. J Orthop Sports Phys Ther. 2003 Sep;33(9):502-12. doi: 10.2519/jospt.2003.33.9.502. PMID 14524509